CLINICAL TRIAL: NCT06026202
Title: Non-Eosinophilic Biological Effects of Interleukin 5 (IL-5) - Role of IL-5 in Suppressing Anti-Viral Immunity in Bronchial Epithelial Cells and Dendritic Cells in Asthma
Brief Title: Non-Eosinophilic Biological Effects of IL-5
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 326910
Record Dates: First submitted 2023-08-25; First posted 2023-09-07 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Asthma
Keywords: Interleukin 5; Bronchial epithelial cells; Peripheral blood mononuclear cells; Peripheral dendritic cells; Interferon; Rhinovirus
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells Bronchial epithelial cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the role of IL-5 in suppressing anti-viral immune responses in bronchial epithelial cells (BECs) and in peripheral blood mononuclear cells (PBMCs) from 5 people with asthma.

DETAILED DESCRIPTION:
IL-5 has been shown to be present in higher levels in those with asthma, more so during viral infection. The investigators know from existing evidence that having increased levels of interferon (IFN) reduces asthma exacerbations and viral load. The investigators suspect that IL-5 reduces the immune response during viral infection in bronchial epithelial cells (BECs) and peripheral blood mononuclear cells (PBMCs) by reducing levels of IFN. The aim is to investigate if increased IL-5 in stable eosinophilic asthma and asthma exacerbations suppresses anti-viral immunity in bronchial epithelial cells and in peripheral blood mononuclear cells directly via IL-5 receptor signalling, suppressing rhinovirus induction of IFNs. The investigators also will evaluate if anti-IL-5 therapies suppress IL-5 concentrations in stable and exacerbated asthma in vivo and whether suppression of IL-5 in vivo restores deficient anti-viral immunity in BECs and PBMCs, thereby protecting against asthma exacerbations.

ELIGIBILITY:
Must be eligible for the study 'Mechanisms of Adverse Effects of Long-Acting Beta-Agonists in Asthma' (MAELABA) (19SM5101).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those with mild asthma on as required salbutamol only.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
IL-5 suppresses anti-viral immunity in BECs and in PBMCs/pDCs directly via IL-5 receptor signalling suppressing RV induction of IFNs. | 1 year
  Expression of IL-5RA, CSF2RB and IFN mRNA and protein in BECs and PBMCs will be measured at baseline and following rhinovirus infection.Viral load will be measured by PCR(copies/ml) of viral RNA in cell lysates and virus release into supernatants by TCID50 assay to determine whether IL-5 augments virus replication.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom